CLINICAL TRIAL: NCT00674466
Title: A Randomized, Double-blind, Placebo-controlled, Multiple-dose, Phase II Study to Evaluate the Efficacy and Safety of 3 Months of Twice-a-week Injections of CJC-1134-PC in Patients With Type 2 Diabetes Mellitus on Metformin Monotherapy
Brief Title: A Study to Evaluate the Efficacy and Safety of CJC-1134-PC in Patients With Type 2 Diabetes Who Are Currently on Metformin Monotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ConjuChem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DM200-102
Record Dates: First submitted 2008-04-18; First posted 2008-05-07 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: GLP-1, incretin, type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Twice-a-week dose of 1.5 mg CJC-1134-PC
  Interventions: Drug: 1.5 mg or 2.0 mg CJC-1134-PC
- 2 (Experimental): Twice-a-week dose of 1.5 mg CJC-1134-PC for 4 weeks, then once-a-week dose of 2.0 mg CJC-1134-PC plus mid-week dosing of placebo
  Interventions: Drug: 1.5 mg or 2.0 mg CJC-1134-PC
- 3 (Placebo Comparator): Twice-a-week placebo for CJC-1134-PC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1.5 mg or 2.0 mg CJC-1134-PC — twice-a-week
  Arms: 1; 2
Drug: Placebo — twice-a-week
  Arms: 3

SUMMARY:
This is a multicenter, randomized, placebo-controlled, double-blind, Phase II study. The objective of this study is to evaluate the efficacy and safety of 12 weeks of treatment with CJC-1134-PC in patients who are currently on metformin monotherapy.

ELIGIBILITY:
Major Inclusion Criteria:

* BMI: 27 to 45 kg/m2
* Stable Type 2 diabetes mellitus for at least 3 months, as defined by the Investigator
* Stable life-style, i.e. diet & physical activity, as determined by the Investigator
* Stable metformin daily dose ≥1000 mg for at least 3 months
* Glycosylated hemoglobin (HbA1c) at screening ≥ 7.1% and ≤ 11%

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Wang, MD, Study Director — ConjuChem Biotechnologies Inc.
Locations (1):
- Maggie Wang, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.5 mg CJC-1134-PC: Twice-a-week dose of 1.5 mg CJC-1134-PC
  1.5 mg CJC-1134-PC: twice-a-week
- 1.5 mg or 2.0 mg CJC-1134-PC: Twice-a-week dose of 1.5 mg CJC-1134-PC for 4 weeks, then once-a-week dose of 2.0 mg CJC-1134-PC plus mid-week dosing of placebo
  1.5 mg or 2.0 mg CJC-1134-PC: twice-a-week
- Placebo: Twice-a-week placebo for CJC-1134-PC
  Placebo: twice-a-week
Period: Overall Study
Arm/Group | 1.5 mg CJC-1134-PC | 1.5 mg or 2.0 mg CJC-1134-PC | Placebo
Started | 30 | 30 | 30
Completed | 23 | 22 | 21
Not Completed | 7 | 8 | 9

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.5 mg CJC-1134-PC | 1.5 mg or 2.0 mg CJC-1134-PC | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 29 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (8.05) | 55.5 (11.06) | 55.2 (8.26) | 55.7 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 19 | 49
  Male | 17 | 13 | 10 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 9 | 27
  Not Hispanic or Latino | 22 | 20 | 20 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 3 | 11
  White | 25 | 23 | 26 | 74
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Reduction of HbA1c From Baseline
Description: Change from baseline
Time Frame: Screening and Day 85
Population: Modified Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Percent (%)
Arm/Group | 1.5 mg CJC-1134-PC | 1.5 mg or 2.0 mg CJC-1134-PC | Placebo
Number analyzed (Participants) | 27 | 27 | 26
Percent (%) | -1.29 (1.226) | -0.55 (0.672) | -0.34 (0.697)

2. Secondary Outcome: Reduction in Fasting Plasma Glucose From Baseline
Description: Change from baseline
Time Frame: Screening and Day 85
Population: Modified Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 1.5 mg CJC-1134-PC | 1.5 mg or 2.0 mg CJC-1134-PC | Placebo
Number analyzed (Participants) | 27 | 27 | 26
mg/dL | -5.88 (62.369) | 4.12 (46.803) | 12.12 (33.210)

3. Secondary Outcome: Reduction in Fasting Body Weight From Baseline
Description: Change from baseline
Time Frame: Screening and Day 85
Population: Modified Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 1.5 mg CJC-1134-PC | 1.5 mg or 2.0 mg CJC-1134-PC | Placebo
Number analyzed (Participants) | 27 | 27 | 26
kg | -1.17 (1.976) | -0.90 (1.873) | -0.39 (2.467)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | 1.5 mg CJC-1134-PC | 1.5 mg or 2.0 mg CJC-1134-PC | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30 | 1/29
Other Adverse Events (participants affected / at risk) | 18/30 | 19/30 | 20/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1.5 mg CJC-1134-PC (N=30) | 1.5 mg or 2.0 mg CJC-1134-PC (N=30) | Placebo (N=29)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Eye infection staphylococcal (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1.5 mg CJC-1134-PC (N=30) | 1.5 mg or 2.0 mg CJC-1134-PC (N=30) | Placebo (N=29)
Nausea (Gastrointestinal disorders) | 8 | 7 | 4
Vomiting (Gastrointestinal disorders) | 7 | 5 | 5
Diarrhea (Gastrointestinal disorders) | 3 | 4 | 6
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 2
Constipation (Gastrointestinal disorders) | 3 | 1 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 8 | 9 | 7
Dizziness (Nervous system disorders) | 3 | 2 | 2
Injection site reaction (General disorders) | 2 | 4 | 3
Fatigue (General disorders) | 4 | 3 | 1
Edema peripheral (General disorders) | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 2 | 3 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes